CLINICAL TRIAL: NCT05706090
Title: Effect of Neurostimulator Usage on Block Success in Costoclavicular Block: a Randomized Controlled Trial
Brief Title: Effect of Neurostimulator Usage on Block Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Döndü Genc Moralar, Associate Professor, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Neurostimulator Usage
Record Dates: First submitted 2022-12-20; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: PATIENTS WITH UPPER EXTREMITY SURGERY
Keywords: Brachial Plexus Block; Nerve Block; Ultrasonography
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group USP (Experimental): The group using ultrasound and injection pressure manometer was named USP
  Interventions: Drug: fentanyl will be added; Procedure: general anesthesia
- Group USPN (Experimental): The group using ultrasound , injection pressure manometer , and neurostimulator was named USPN
  Interventions: Drug: fentanyl will be added; Procedure: general anesthesia

INTERVENTIONS:
Drug: fentanyl will be added — If adequate anagesia is not provided with the block, 1 microgram/kg of fentanyl will be added
Procedure: general anesthesia — If adequate anagesia is not provided with the block, general anesthesia will be administered.

SUMMARY:
The need of a neurostimulator for a successful nerve block was questioned in different block types after ultrasound has become standard. The aim of this clinical study was to determine the effect of neurostimulator use on block success in costoclavicular block

ELIGIBILITY:
Inclusion Criteria:

* Class I, II and III of American Society of Anesthesiologists (ASA) classification
* being between 18 and 80 years of age,
* body mass index (BMI) between 18 and 35 kg/m2

Exclusion Criteria:

* Patients who did not give consent,
* were above ASA III,
* pregnant,
* had a neuromuscular disease,
* bleeding diathesis,
* a local anesthetic allergy,
* an infection in the area where nerve block would be applied, and
* had previously operated from the infraclavicular fossa were not included in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
The block success rate (ratio of successful blocks to all blocks) | during procedure
  The block was considered unsuccessful in case of analgesic need during the surgery or transition to general anesthesia, otherwise, these patients were included in the successful block group.

SECONDARY OUTCOMES:
Block application time | 30 minutes
  THE TIME BETWEEN THE NEEDLE ENTRY THROUGH THE SKIN AND THE OUTPUT OF THE NEEDLE AFTER LOCAL ANESTHETICS IS GIVEN, WAS RECORDED AS THE APPLICATION TIME
time to readiness for surgery | 30 minutes
  Sensory and motor block levels were evaluated in the median, radial, ulnar and musculocutaneous nerve traces at 5-minute intervals for 30 minutes. An ice pack was used for sensory block evaluation. It was scored as follows; 0: completely felt; 1: has a sense of touch; no cold; 2: no sense of touch. Lateral surface of the forearm for the musculocutaneous nerve, the surface of the thumb facing the palm for the median nerve, the inner surface of the 5th finger for the ulnar nerve, and the posterior surface of the hand for the radial nerve were used for sensorial evaluation. Motor block was scored as follows; 0: full motion; 1: paresis; 2: complete block. Elbow flexion for the musculocutaneous nerve, thumb opposition for the median nerve, 5th finger abduction for the ulnar nerve, and wrist extension for the radial nerve were used to evaluate motor block. The block was considered successful if the total score was 14 or higher, with a total sensory score of at least 7.
number of needle passes | 30 minutes
  . The number of needle passes was calculated by adding each needle advancement exceeding 10 mm to the first needle insertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazoosmanpasa Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No